CLINICAL TRIAL: NCT06651151
Title: NeoLIPA: a Single Center Phase II Open Label Study of Neoadjuvant LTX-315 in Combination with Pembrolizumab in Patients with Clinically Detectable and Resectable Stage III-IV Melanoma
Brief Title: NeoLIPA: Neoadjuvant LTX-315 in Combination with Pembrolizumab in Resectable Stage III/IV Melanoma
Acronym: NeoLIPA
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: Lytix Biopharma AS (Industry)
Responsible Party: Principal Investigator, Henrik Jespersen, Head of Melanoma Oncology, Group Leader Melanoma Research, Oslo University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023_16; 2023-508649-42-00 (EU CTIS Number)
Record Dates: First submitted 2024-10-18; First posted 2024-10-21 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: Melanoma Stage IIIB-IV
Keywords: Melanoma; Neoadjuvant; Pembrolizumab; Oncolytic peptide
MeSH Terms: conditions — Melanoma | interventions — LTX-315; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental (Experimental): LTX-315 will be injected directly into the selected tumor once weekly for a maximum of 5 dosing days.
  Pembrolizumab will be given as 200 mg IV infusion over 30 minutes every 3 weeks for a maximum of 18 doses of which three doses will be given prior to the planned surgery.
  Interventions: Drug: LTX-315 + pembrolizumab

INTERVENTIONS:
Drug: LTX-315 + pembrolizumab — LTX-315 as intratumoral injection once weekly for a maximum of 5 dosing days, in combination with pembrolizumab as intravenous infusion, 200 mg every 3 weeks for a maximum of 18 doses

SUMMARY:
This clinical trial aims to evaluate the effectiveness of a new treatment approach for patients with stage III or IV melanoma that has spread to other parts of the body but can still be surgically removed. The study combines two treatments: LTX-315 and pembrolizumab.

Melanoma that has spread to other parts of the body can often be treated with surgery. Despite surgery, there is a high risk of the cancer coming back. Pembrolizumab, an immune checkpoint inhibitor, can reduce this risk when given after surgery. Recent studies have shown that giving pembrolizumab before surgery, along with post-surgery treatment, might be more effective than giving it only after surgery. However, many patients still experience cancer recurrence. Combining pembrolizumab with LTX-315, which triggers a different immune response, might improve the treatment&#39;s effectiveness and reduce the risk of cancer progression before surgery.

This is an open-label Phase II study, meaning both the researchers and participants will know which treatments are being given. The study will be conducted at a single center and will involve about 27 participants. They will receive LTX-315 and pembrolizumab before their planned surgery to see if this combination could be more effective than pembrolizumab alone.

The primary goal is to assess the tumors response to the neoadjuvant (pre-surgery) treatment, specifically looking at the rate of pathological complete response (pCR), where no cancer is detected in the removed tumor tissue.

DETAILED DESCRIPTION:
This is a single arm, single center, open-label phase II study to assess the effect of neoadjuvant LTX-315 in combination with pembrolizumab in patients with clinically detectable and resectable stage III-IV melanoma.

Clinically detectable, fully resectable stage III or oligometastatic IV melanoma can be cured with surgery but has a very high risk of local or systemic recurrence. The risk of recurrence can be significantly reduced by adjuvant treatment with a PD-1 inhibitor. Due to the mode of action of PD-1 inhibitors (stimulating tumor reactive T cells), there is reason to believe that their effect is enhanced if given before definitive surgery and removal of tumor reactive T cells in the tumor microenvironment. Indeed, it was recently shown that the effect is greatly improved if three doses of pembrolizumab are administered prior to surgery (neoadjuvant), followed by 15 doses in the adjuvant setting, compared to giving 18 doses adjuvant.

Several studies have shown that pathologic complete response (pCR) after neoadjuvant treatment correlates with recurrence-free survival (RFS). The pCR rate neoadjuvant pembrolizumab is only modest (20%), and for 8% of the patients, disease progression in the neoadjuvant phase precludes the planned surgery.

LTX-315 is an oncolytic peptide generated from a host defense peptide and has both a direct killing activity and immunomodulatory properties. By inducing cell lysis and immunogenic cell death, LTX-315 can lead to increased T-cell infiltration, broadened repertoire of tumor antigens and increased diversity of T-cell clones, and thus has the potential to enhance the effect of pembrolizumab. Furthermore, the addition of LTX-315 to neoadjuvant pembrolizumab can lower risk of disease progression precluding surgery.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be 18 years of age inclusive, at the time of signing the informed consent.
* Histologically confirmed, clinically detectable stage III-IV(M1a) melanoma, judged fully resectable and eligible for neoadjuvant treatment by consensus at a multidisciplinary tumor board. Patients with melanoma of cutaneous (including acral) or mucosal (including conjunctival) origin are eligible. Clinically detectable is defined as being apparent and measurable by radiological assessments or physical examination.
* Measurable disease as per RECIST version 1.1 criteria.
* Judged medically fit to undergo the planned surgery by the surgical team.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Have at least one superficial cutaneous, subcutaneous or lymph node lesion available for injection with a maximum mean longest perpendicular diameter (LPD) of 3.0 cm.
* Willing to undergo an additional tumor biopsy and submit biopsy and surgical specimens
* Adequate organ function as defined below:

  1. Hemoglobin > 9 g/dL
  2. Absolute neutrophil count (ANC) ≥ 1.0 x 109/L
  3. Platelet count ≥ 80 x 109/L

  e. Serum bilirubin ≤ 1.5 x institutional upper limit of normal (ULN) f. AST and ALT ≤2.5 x ULN g. Albumin >30 g/L h. Serum creatinine ≤1.5 X ULN OR measured creatinine clearance (CL) >30 mL/min
* Female participants are willing to use contraceptive measures as prescribed by the protocol from study visit 1 to 120 days after the last dose of study intervention. Women of childbearing potential must have a negative urine or serum pregnancy test within 72 hours of first study intervention.
* Capable of giving signed informed consent as described in section 10.1 which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.

Exclusion Criteria:

* Uveal melanoma. Patients with acral, mucosal or conjunctival melanoma are eligible.
* History of brain, bone, liver metastases or leptomeningeal metastases.
* Patients with stage IV disease having ≥4 metastatic sites.
* A history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating Investigator.
* Active autoimmune disease requiring systemic immunomodulatory treatment. Replacement therapy (e.g. physiologic doses of corticosteroids, insulin, thyroxine) is allowed.
* Patient has history of, or any evidence of interstitial lung disease (ILD) or non-infectious pneumonitis that required systemic corticosteroids.
* Prior malignancy that require concurrent therapy.
* Allergy/hypersensitivity to prophylactic treatments; known hypersensitivity to pembrolizumab or LTX-315 or any of their excipients
* Previous treatment with anti-cancer immunotherapy, including (but not limited to) CTLA-4 or PD-1 inhibitors. Prior non-immunotherapy adjuvant treatment (e.g.

dabrafenib + trametinib or radiotherapy), and regional therapy such as ECT or ILP is permitted (≥ 12 weeks prior to enrollment).

* Currently taking immunosuppressive agents or use of systemic corticosteroids (≥10 mg of prednisolone or equivalent) or other systemic immunosuppressive drugs within 28 days prior to study drug administration. Topical and inhaled corticosteroids are allowed.
* Have received a live vaccine within 30 days prior to first dose of treatment
* Have received an investigational drug within 4 weeks to day 1, or are scheduled to receive one during the treatment period.
* Pregnant or breastfeeding.
* Any reason why, in the opinion of the investigator, the patient should not participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2031-05 (Estimated)

PRIMARY OUTCOMES:
Complete Pathologic Response Rate | 12 weeks after start of treatment
  Rate of pathologic complete response (pCR), defined as complete absence of viable tumor in the treated tumor bed.

SECONDARY OUTCOMES:
Safety Evaluation | Continously from first dose of treatment to 90 days after last study drug administration
  Frequency, nature and severity of AE according to NCI CTCAE v 5.0:
  * All AEs
  * LTX-315 treatment-related AEs
  * LTX-315 and/or pembrolizumab treatment-related AEs
Objective response rate (ORR) | After 12 weeks of treatment
  Rate of CR or PR as per RECIST version 1.1 prior to surgery
Pathologic Response Rate | After 12 weeks of treatment
  Rate of partial (less than 50% of the treated tumor bed is occupied by viable tumor cell) or complete pathologic response.
  Rate of Major Pathologic Response (MPR) defined as complete or near-complete (less than 10% of viable tumor in the treated tumor bed) pathologic response
Event free survival (EFS) | From first dose of treatment to two years
  Defined as time from start of treatment to progression of disease that precludes surgery, recurrence (local or distant) or death
Recurrence free survival (RFS) | Two years after surgery
  Defined as the time from surgery to recurrence or death.
Overall Survival (OS) | Three years after surgery
  Overall Survival
Quality of Life (QoL) | From first dose to end of treatment at approximately 1.5 years
  Patient reported outcomes (PRO)

CONTACTS AND LOCATIONS:
Locations (1):
- Oslo University Hospital, Oslo, Oslo County, Norway